CLINICAL TRIAL: NCT06342349
Title: A Randomized, Double-blind, Controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of the Quadrivalent Influenza Virus Split Vaccine (MDCK Cells) for Individuals Aged 6 Months and Above.
Brief Title: A Clinical Trial of Quadrivalent Influenza Virus Split Vaccine (MDCK Cells) for Individuals Aged 6 Months and Above.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-V03-I
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Influenza
Keywords: Quadrivalent influenza virus split vaccine; MDCK cells; Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: This is a single center, randomized, double-blind, controlled phase I clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SIBP-V03-I (Experimental): Quadrivalent influenza virus split vaccine (MDCK cells)
  Interventions: Biological: Quadrivalent influenza virus split vaccine (MDCK cells)
- QTV (chicken embryo) (Active Comparator): Quadrivalent influenza virus split vaccine (chicken embryo)
  Interventions: Biological: Quadrivalent influenza virus split vaccine (Chicken embryo)
- Placebo (Placebo Comparator): Phosphate buffer solution
  Interventions: Other: Phosphate buffer solution

INTERVENTIONS:
Biological: Quadrivalent influenza virus split vaccine (MDCK cells) — Quadrivalent influenza vaccine made from cell matrix (0.5ml/dose).
  Arms: SIBP-V03-I
Biological: Quadrivalent influenza virus split vaccine (Chicken embryo) — Quadrivalent influenza vaccine made from chicken embryo(0.5ml/dose).
  Arms: QTV (chicken embryo)
Other: Phosphate buffer solution — Phosphate buffer solution without vaccine antigen(0.5ml/dose).
  Arms: Placebo

SUMMARY:
To evaluate the safety of administering 1 or 2 doses of the quadrivalent influenza virus split vaccine (MDCK cells) (0.5ml/dose) in individuals aged 6 months and above.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, controlled phase I clinical trial. Plan to include 300 participants aged 6 months and above. The experiment was divided into 5 age groups, with 60 cases each aged 6-35 months, 3-8 years, 9-17 years, 18-59 years, and ≥ 60 years old. Each age group was randomly assigned to the experimental group, control group, or placebo group in a 1:1:1 ratio. Among them, the participants aged 6 to 35 months and 3 to 8 years old will receive 2 doses throughout the entire process, with an interval of 28 days between each dose. Participants aged 9-17, 18-59, and ≥ 60 years old are vaccinated with one dose throughout the entire process.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 6 months or more on the day of enrollment who can provide legal identification documents.
* Volunteers and/or their legal guardians (or entrusted persons) have informed consent, voluntarily participate, and sign an informed consent form.
* Volunteers and/or their legal guardians (or entrusted persons) have the ability (non-illiterate) to understand the research procedures, could use thermometers, scales, and fill out diary cards as required, and can comply with the requirements of the clinical trial protocol to complete the clinical study.

Exclusion Criteria:

（Exclusion criteria for the first dose）

* On the day of enrollment, the underarm temperature of individuals ≤ 14 years old is ≥ 37.5 ℃, and on the day of enrollment, the underarm temperature of individuals>14 years old is ≥ 37.3 ℃.
* Women of childbearing age (from menarche to menopause for ≤ 1 year) who have tested positive for urinary pregnancy test, and those who are breastfeeding, pregnant, or planning to conceive within 6 months.
* Have had or are currently suffering from influenza within the past 3 months (confirmed by clinical, serological, or microbiological methods).
* Individuals aged 6 months to 8 years have previously received any influenza vaccine (including registered or experimental) or have planned to receive any influenza vaccine during the study period. Individuals aged 9 and above have received any influenza vaccine (including registered or experimental) within the past 6 months or have planned to receive any influenza vaccine within the past 6 months.

Has a history of allergic reactions to any component of the research vaccine, including consuming eggs or using gentamicin sulfate.

* Has any history of severe allergies to vaccines or drugs in the past. Population aged 6 to 35 months: premature birth (delivered before the 37th week of pregnancy), low birth weight (birth weight<2500g) infants.
* Population aged 6 to 35 months: those with a history of difficult childbirth, suffocation rescue, and neurological damage.
* Congenital malformations (clinically significant according to researchers) or developmental disorders, genetic defects, and severe malnutrition.
* Population aged 3-8 years and 6-35 months: individuals with abnormal growth and development, severe eczema.
* Suffering from acute illness or being in the acute phase of chronic illness within 3 days before vaccination.
* Used antipyretic and analgesic drugs or anti allergic drugs within 3 days before vaccination.
* Suffering from serious chronic diseases, serious cardiovascular diseases, hypertension beyond drug control (systolic pressure ≥ 140mmHg or diastolic pressure ≥ 90mmHg, only applicable to people aged 18 and above), diabetes with complications, liver and kidney diseases, malignant tumors, etc.
* Have a history of receiving attenuated live vaccines within 14 days (including the 14th day) before vaccination and have a history of receiving other vaccines within 7 days (including the 7th day).
* Individuals who receive immunotherapy or immunosuppressive therapy within 3 months (continuous oral or intravenous for more than 14 days).
* Suffering from congenital or acquired immunodeficiency, human immunodeficiency virus infection, lymphoma, leukemia, or other autoimmune diseases.
* Asthma history, unstable in the past two years requiring emergency treatment, hospitalization, intubation, oral or intravenous corticosteroids.
* Have received blood or blood related products within the past 6 months.
* Individuals with progressive neurological disorders have a history of seizures, epilepsy, encephalopathy, Guillain Barre syndrome, psychiatric disorders, transverse myelitis, or family history.
* Have a history of abnormal coagulation function (such as coagulation factor deficiency, coagulation related diseases), or use anticoagulants within 3 weeks before vaccination.
* Non splenic, functional non splenic, splenectomy, or partial resection of other important organs.
* Plan to relocate before the end of the study or leave the local area for a long time during the scheduled study visit period.
* Being or planning to participate in other clinical trials in the near future.
* Abnormal laboratory testing indicators, except for minor abnormalities judged by doctors to have no clinical significance.
* The researcher determines any situation that is not suitable for participation in this clinical trial.

（Exclusion criteria for the second dose）

* On the day of vaccination, the axillary body temperature is ≥ 37.5 ℃.
* Fever (axillary temperature ≥ 38.5 ℃) within 3 days before vaccination, or use of antipyretic and analgesic drugs or anti allergic drugs within 3 days before vaccination.
* Suffering from various acute or chronic diseases with acute attacks within 3 days before vaccination.
* Insufficient interval between vaccination of other vaccines (with a history of receiving attenuated live vaccines within 14 days (including the 14th day) before vaccination, and a history of receiving other vaccines within 7 days (including the 7th day).
* Other situations where researchers believe vaccination should be postponed.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Solicited Adverse Events (AEs) | 7 days after each dose of vaccination
  Adverse events defined by the protocol that occurred to the participant during 0-7 days after each dose of vaccination.
Unsolicited Adverse Events | 28 or 30 days after each dose of vaccination
  Other adverse events that occurred among participants within 0-28/30 days after each vaccination, in addition to the solicited adverse events.
Serious Adverse Events (SAE) | 6 months after the last dose
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.

SECONDARY OUTCOMES:
Seroconversion rate | 30 days after the last dose of vaccination
  30 days after the full vaccination of all participants with the experimental vaccine or control vaccine, the HI antibody seroconversion rate against any subtype of influenza virus in the experimental vaccine group and the control vaccine group.
Ratio of ≥1:40 | 30 days after the last dose of vaccination
  30 days after the full vaccination of all participants with the experimental vaccine or control vaccine, the ratio of HI antibody titers ≥ 1:40 against any subtype of influenza virus in the experimental vaccine group and the control vaccine group.
Geometric mean increase (GMI) | 30 days after the last dose of vaccination
  30 days after the full vaccination of all participants with the experimental vaccine or control vaccine, GMI of HI antibodies against any subtype of influenza virus in the experimental vaccine group and the control vaccine group.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Li, Principal Investigator — 0351-7553168
Locations (1):
- Shanxi Provincial Center for Disease Prevention and Control, Shanxi, China

IPD SHARING:
Plan to Share IPD: No